CLINICAL TRIAL: NCT00327951
Title: The Impact of Weight Gain in the Pre-operative Infant With Trisomy 21 (Down Syndrome) and Complete Atrioventricular Canal (CAVC)
Brief Title: Infant Weight Gain With Trisomy 21 and CAVC
Status: Terminated | Type: Observational
Why Stopped: sufficient data collected for significant conclusion
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Children's Healthcare of Atlanta Institutional Review Board, IRB Chairman
Other Study IDs: 06-109
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2008-02

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; weight gain pre-operative; trisomy 21; complete atrioventricular canal
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Down Syndrome; Complete atrioventricular septal defect

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Failure to thrive and difficulty gaining weight is a sign of uncompensated congestive heart failure (CHF). Infants with Trisomy 21 and complete atrioventricular canal defects (CAVC) frequently develop uncompensated CHF and weight gain failure pre-operatively. A weight of 5 kg has been suggested as optimal for timing of CAVC repair. A delay in surgical repair often occurs if weight gain stalls and reaches a plateau prior to reaching 5 kg. A retrospective review performed by Kogon, et al, of children undergoing surgery for VSD at CHOA at Egleston recently reported that age and weight at surgery may not, however, be associated with adverse surgical outcome.

The purpose of this study is to determine the optimal timing for surgical correction of CAVC in Trisomy 21 infants based on reaching a plateau of failed weight gain despite maximal anti-congestive and nutritional therapy.

DETAILED DESCRIPTION:
A retrospective chart review of 100 infants with Trisomy 21 and CAVC operated at CHOA at Egleston between January 1, 2001 and March 24, 2006 will be performed. Graphs of birth weight and rate of weight gain over time will be plotted for each patient and for the group as a whole. The point of reaching a plateau of weight gain will be decided for each patient and indexed for birth weight. Medical management will be detailed, i.e. all medications and all dietary information (caloric density of formula, route of administration). This medical management will be indexed as a function on the weight gain chart. Medical complications (such as respiratory infections, gastroenteritis, hospitalizations, and additional non-cardiac medications) will likewise be plotted and segmented according to position relative to the weight gain plateau. Age at eventual surgery and whether surgical date was delayed by complications will be noted. Surgical cardiopulmonary bypass time and morbidity and mortality will be noted. Postoperative length of ventilator support, length of stay in the CICU and total length of stay will be determined and also displayed as a function of body weight and as a function of time at plateau weight. Postoperative morbidity and mortality for the three months after repair will be noted, including all cause hospital re-admissions and outpatient medical complications (such as respiratory infections, gastroenteritis, and the need for continued medications for CHF).

ELIGIBILITY:
Inclusion Criteria:

* Infants with Trisomy 21 and CAVC operated on at CHOA at Egleston between January 1, 2001 and December 31, 2005 will be included in the study.

Exclusion Criteria:

* Patients will be excluded if the following information is not available:

A. Birth weight B. Weight at operation C. Incomplete medical records e.g. patient followed preoperatively elsewhere

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients' charts from Children's Healthcare of Atlanta
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2001-01; Primary Completion 2006-03 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy M Alderson, MD, Principal Investigator — Emory University @ Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States